CLINICAL TRIAL: NCT05327829
Title: Stimulating After Recovery From Traumatic Brain Injury
Acronym: SMART
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-FY2023-678
Record Dates: First submitted 2022-02-28; First posted 2022-04-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Block design
Who Masked: Participant
Masking Description: Participants are blinded to stimulation versus no stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham (Sham Comparator): No stimulation
  Interventions: Behavioral: COGED
- Stimulation (Active Comparator): Stimulation
  Interventions: Combination Product: External non-invasive stimulation; Behavioral: COGED

INTERVENTIONS:
Combination Product: External non-invasive stimulation — The participants are randomized into the block design of sham or tACS during the first three appointments or the last three appointments. Eye tracking will be used to test the predominant focus of decisions during the gaze phase on costs or difficulty levels during the COGED. The study is investigating the use of neuromodulation after TBI for improved cognitive function.
  Arms: Stimulation
Behavioral: COGED — The COGED task consists of the classic N-back task of working memory-based decision making, followed by a valuation phase. The N-back phase of the task allows calculation of cognitive performance of a working memory task. During valuation, participants receive titrating offers of differing amounts of money to perform different difficulty levels of the N-back. The result is an effort discounting curve used to measure the individual effort cost. Effort discounting curves show the perceived cognitive effort required to complete each level of the task relative to another (typically the 1-back).

SUMMARY:
This is a preliminary, prospective interventional study to investigate the feasibility of using transcutaneous alternating current stimulation (TACS) after a traumatic brain injury (TBI) to improve cognitive function and decision-making.

DETAILED DESCRIPTION:
All participants engaged in the study will participate once weekly for six weeks at Hennepin Healthcare Systems, Inc. (HHS). Each participant will be randomized into the block design of sham or tACS during the first three appointments or the last three appointments. While participating, both the tACS will be applied in accordance with the manufacturer's suggested use. Participants will complete computer-based tasks, while taking part in either the sham or tACS stimulation. The study is investigating the use of neuromodulation after Traumatic Brain Injury (TBI) for improved cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Diagnosis of a mild to moderate TBI (GCS > 8 on admission)
* Able to perform a computerized assessment
* Willing to attend all scheduled appointments
* Able to undergo the informed consent process

Healthy participants:

* Adults 18 years and older
* Able to perform a computerized assessment
* Willing to attend all scheduled appointments
* Able to undergo the informed consent process

Exclusion Criteria:

* Open wound on scalp
* Severe TBI diagnosis or GCS of less than 8 on admission
* Non-English speaking
* Incarcerated
* Implanted defibrillator or pacemaker
* Visual impairment that hinders ability to complete computerized assessments

Healthy subject exclusion criteria:

* Less than 18 years of age
* Open wound on scalp
* TBI diagnosis
* Non-English speaking
* Incarcerated
* Implanted defibrillator or pacemaker
* Visual impairment that hinders ability to complete computerized assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using non-invasive stimulation to improve Cognitive Flexibility after TBI | 3 years
  Using non-invasive transcranial alternating current stimulation, it will be determined if this study is feasible for improving cognitive recovery after mild to moderate brain injury. To determine the sum total of completion rate of study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No